CLINICAL TRIAL: NCT06287372
Title: Comparison of Changes in Intra-myocardial Amino Acids During Use of Calafiore and Modified Del Nido Cardioplegic Solutions in Routine Coronary Artery Bypass Surgery
Brief Title: Comparison of Changes in Intra-myocardial Amino Acids During Use of Calafiore and Modified Del Nido Cardioplegia
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Principal Investigator, Mohammad Bashar Izzat, Professor, Damascus University
Other Study IDs: 3261
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Myocardial Injury; Cardiac Surgery; Myocardial Protection
Keywords: cardioplegia; coronary artery bypass grafting; amino acid
MeSH Terms: interventions — Cardioplegic Solutions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Calafiore cardioplegia: Patients were randomly assigned to undergo surgery using one of two methods for myocardial protection:
  • Group 1: Calafiore intermittent antegrade warm blood cardioplegia (consisting of normothermic pump blood, potassium chloride 2 mEq/ml and magnesium sulfate 50%). This cardioplegic solution was administered at 37 degrees C following application of the aortic cross-clamp and repeated after completion of each distal coronary anastomosis as described previously.
  Interventions: Other: Cardioplegic solution
- Group 2: del Nido cardioplegia: • Group 2: Modified del Nido intermittent antegrade cold blood cardioplegic solution (consisting of 750 ml of lactated Ringer solution, 200 ml of pump blood, 13 ml of sodium bicarbonate 8.4%, 16 ml of mannitol 20%, 4 ml of magnesium sulfate 50%, 13 ml of lidocaine 2% and 13 ml of potassium chloride 2 mEq/ml). This solution was administered as a 1-liter bolus at 3-4 degrees C following application of the aortic cross-clamp, and repeated as a 500 ml bolus if cross-clamp time extended beyond 60 minutes (none of the patients in this study).
  Interventions: Other: Cardioplegic solution

INTERVENTIONS:
Other: Cardioplegic solution — Patients were randomly assigned to undergo surgery using one of two methods for myocardial protection

SUMMARY:
The aim of the present study was to investigate intra-operative changes in markers of myocardial injury and myocardial intracellular amino acids during ischemia and reperfusion, comparing two methods of myocardial protection; Calafiore intermittent antegrade warm blood cardioplegia or modified del Nido intermittent antegrade cold blood cardioplegia in routine coronary artery bypass grafting procedures.

DETAILED DESCRIPTION:
Twenty consecutive patients undergoing elective primary coronary artery bypass grafting were enrolled in this study. Patients were excluded from this study if they had suffered from previous myocardial infarction, had reduced ejection fraction or were undergoing combined or repeated surgery. Patients were randomly assigned to undergo surgery using one of two methods for myocardial protection:

* Group 1: Calafiore intermittent antegrade warm blood cardioplegia (consisting of normothermic pump blood, potassium chloride 2 mEq/ml and magnesium sulfate 50%). This cardioplegic solution was administered at 37 degrees C following application of the aortic cross-clamp and repeated after completion of each distal coronary anastomosis as described previously.
* Group 2: Modified del Nido intermittent antegrade cold blood cardioplegic solution (consisting of 750 ml of lactated Ringer solution, 200 ml of pump blood, 13 ml of sodium bicarbonate 8.4%, 16 ml of mannitol 20%, 4 ml of magnesium sulfate 50%, 13 ml of lidocaine 2% and 13 ml of potassium chloride 2 mEq/ml). This solution was administered as a 1-liter bolus at 3-4 degrees C following application of the aortic cross-clamp, and repeated as a 500 ml bolus if cross-clamp time extended beyond 60 minutes (none of the patients in this study).

Each patient enrolled in the study gave a written informed consent for the publication of the study data, and the study protocol conformed to the ethical guidelines of the 1975 Declaration of Helsinki as reflected in a priori approval by the local human research committee number 171 dated 13 April 2022

Collection of blood samples and myocardial biopsies Peripheral blood samples were collected immediately prior to surgery and at 4, 12, 24 and 48 hours postoperatively and were used for determination of blood concentrations of cardiac enzymes (CK-MB and troponin I).

Myocardial biopsies (4-14 mg wet weight) were taken using a Tru-cut needle from the apex of the left ventricle in every patient as follows:

* Biopsy 1: "Resting specimen", immediately after beginning of extracorporeal circulation.
* Biopsy 2: "Ischemic specimen", 30 minutes after application of the aortic cross-clamp.
* Biopsy 3: "Reperfusion specimen", 20 minutes following the removal of aortic cross-clamp.

Each specimen was immediately snap-frozen in liquid nitrogen (-185 degrees C) until processing for the analyses of amino acids and lactic acid.

Determination of cardiac enzymes (CK-MB and troponin I) Analyses were carried out using an immunofluorescence scanner (iChroma II, Boditech Med Incorporated, Korea and Obelis s.a, Belgium). Blood levels of CK-MB were expressed as mg/dl and levels of troponin I were expressed as ng/ml.

Determination of myocardial amino acid and lactic acid concentrations Each frozen biopsy specimen was weighed (Laboratory Analytical Balance, Sartorius, Germany), crushed in liquid nitrogen and homogenized in 1000 micro mol of 0.9% normal saline. A 400 micro mol sample of the homogenate was transferred to an Eppendorf tube and 100 micro mol of HPLC water was added. Each sample was then stored at 4 degrees C for one hour, after which it was centrifuged at 10000 round/min for 5 minutes. A 400 micro mol sample of the supernatant was filtered through a Vivaspin® 500 membrane filter 0.2 µm (Satorius, Germany), transferred to an Eppendorf tube and was centrifuged at 10000 round/min for 5 minutes. A 300 micro mol sample of the filtrate was transferred to an Eppendorf tube and an equal volume of sample dilution buffer (membraPure, Germany) was added. This solution was used for determining the concentrations of 7 amino acids (alanine, glutamine, glutamic acid, glycine, lysine, ornithine and taurine) using the A300 Amino Acid Analyzer (ARACUS, membraPure, Germany). Lactic acid concentrations were also measured using a dedicated plasma lactate determination kit and analyzer (LACT2, cobas, Roche Diagnostics GmbH, Germany). Concentrations of amino acids and lactic acid were expressed as micro mol/g wet weight.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing elective primary coronary artery bypass grafting were enrolled in this study.

Exclusion Criteria:

* Patients were excluded from this study if they had suffered from previous myocardial infarction, had reduced ejection fraction or were undergoing combined or repeated surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Twenty consecutive patients undergoing elective primary coronary artery bypass grafting were enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Changes in markers of myocardial injury | 4, 12, 24 and 48 hours postoperatively
  Changes in release of myocardial CK-MB and troponin I

SECONDARY OUTCOMES:
Changes in myocardial amino acid concentrations | 2-3 hours
  Changes in myocardial intracellular concentrations of 7 amino acids (alanine, glutamine, glutamic acid, glycine, lysine, ornithine and taurine)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Bashar Izzat, Study Director — Damascus University
Locations (1):
- Damascus University Cardiac Surgery Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided
Data will be uploaded on (figshare) data repository site